CLINICAL TRIAL: NCT00733486
Title: A Prospective, Non-Comparative Study to Evaluate the Performance of the DePuy Low Contact Stress (LCS®) Complete Anterior-Posterior Glide (AP Glide) Mobile Bearing Knee System in Primary Knee Arthroplasty
Brief Title: A Study to Evaluate the Performance of the DePuy Low Contact Stress (LCS®) Complete Anterior-Posterior Glide (APG) Mobile Bearing Knee
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated at 2 years as investigators were unable to continue participation in the study.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT 02/41
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty, Replacement, Knee, LCS Complete APG (MeSH);
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L.C.S. APG Knee Anterior Posterior Glide knee (Other): Orthopaedic implant for primary knee replacement
  Interventions: Device: L.C.S. APG Knee Anterior Posterior Glide knee

INTERVENTIONS:
Device: L.C.S. APG Knee Anterior Posterior Glide knee — Orthopaedic implant for primary knee replacement

SUMMARY:
The primary objective of this investigation is to determine the survivorship of the LCS Complete AP Glide mobile bearing knee prosthesis at 5 years.

The secondary objectives of this investigation are to evaluate the clinical performance of the LCS® Complete AP Glide mobile bearing knee prosthesis and to determine its long-term survivorship.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged between 45 and 85 years inclusive.
* Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
* Subjects who present with any pathology that in the opinion of the clinical investigator requires a primary total knee arthroplasty.
* Subjects who have an intact posterior cruciate ligament and well functioning medial and lateral collateral ligaments.
* Subjects who in the opinion of the Clinical Investigator are considered to be suitable for treatment with the LCS Complete AP Glide mobile bearing knee system, according to the indications specified in the package insert leaflet.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.
* Revision of an existing knee implant (including unicompartmental implants).
* Female subjects who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical study with an investigational product in the last month (30 days).
* Subjects who are currently involved in any personal injury litigation claims.
* Subjects involved in personal Medical-Legal claims.
* Subjects with a known history of poor compliance to medical treatment.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2005-08; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
A survival analysis of the LCS® Complete AP Glide knee prosthesis at five years. | 2 years

SECONDARY OUTCOMES:
Changes from baseline to 3 months post-operative assessment in:Clinical outcome (stability, pain, range of motion and function), using the American Knee Society Score. | Pre-op to 3 months
  American Knee Society (AKS) knee score is a 0-100 point score (where 100 indicates excellent knee condition) that evaluates the affected knee. The knee score is composed of Pain, Range of Motion, and Stability.
  American Knee Society (AKS) function score is a 0-100 point score (where 100 indicates excellent knee function) that evaluates the affected knee
Change from baseline to 1 year post-operative assessment in clinical outcome (stability, pain, range of motion and function) using the American Society Score | Pre-op to 1 year
  American Knee Society (AKS) knee score is a 0-100 point score (where 100 indicates excellent knee condition) that evaluates the affected knee. The knee score is composed of Pain, Range of Motion, and Stability.
  American Knee Society (AKS) function score is a 0-100 point score (where 100 indicates excellent knee function) that evaluates the affected knee
Change from baseline to 3 year post-operative assessment in clinical outcome (stability, pain, range of motion and function) using the American Society Score | Pre-op to 3 years
  American Knee Society (AKS) knee score is a 0-100 point score (where 100 indicates excellent knee condition) that evaluates the affected knee. The knee score is composed of Pain, Range of Motion, and Stability.
  American Knee Society (AKS) function score is a 0-100 point score (where 100 indicates excellent knee function) that evaluates the affected knee
Incidence of anterior knee pain and patellar function using the Patellar Score | 3 months post-operatively
  The Patellar Score is a 1 to 30 point outcome score (where 30 indicates the best outcome) that evaluates the patella of the affected knee. The patellar score is composed of Anterior Knee Pain (max 15 points), Quadriceps Strength (max 5 points), Ability to rise from chair (max 5 points), and Stair-climbing (max 5 points).
Incidence of anterior knee pain and patellar function using the Patellar Score | 1 year post-operatively
  The Patellar Score is a 1 to 30 point outcome score (where 30 indicates the best outcome) that evaluates the patella of the affected knee. The patellar score is composed of Anterior Knee Pain (max 15 points), Quadriceps Strength (max 5 points), Ability to rise from chair (max 5 points), and Stair-climbing (max 5 points).
Incidence of anterior knee pain and patellar function using the Patellar Score | 3 year post-operatively
  The Patellar Score is a 1 to 30 point outcome score (where 30 indicates the best outcome) that evaluates the patella of the affected knee. The patellar score is composed of Anterior Knee Pain (max 15 points), Quadriceps Strength (max 5 points), Ability to rise from chair (max 5 points), and Stair-climbing (max 5 points).
Patient derived outcome in terms of joint specific quality of life, as determined by the Oxford Knee Score | 3 months post-operatively
  The Oxford Knee Score (OKS) is a 12 to 60 point patient reported outcome (PRO) score (where 12 indicates the best outcome) that evaluates the affected knee. The total score is composed of Pain and Function.
Patient derived outcome in terms of joint specific quality of life, as determined by the Oxford Knee Score | 1 year post-operatively
  The Oxford Knee Score (OKS) is a 12 to 60 point patient reported outcome (PRO) score (where 12 indicates the best outcome) that evaluates the affected knee. The total score is composed of Pain and Function.
Patient derived outcome in terms of joint specific quality of life, as determined by the Oxford Knee Score | 3 years post-operatively
  The Oxford Knee Score (OKS) is a 12 to 60 point patient reported outcome (PRO) score (where 12 indicates the best outcome) that evaluates the affected knee. The total score is composed of Pain and Function.
Patient derived outcome in terms of general quality of life, as determined by the SF-12 | 3 months post-operatively
  The 12-Item Short Form Health Survey (SF-12) is a patient reported outcome survey that evaluates functional health and well-being. The survey is converted into 2 summary measures that are scored from 0 to 100 (where 100 indicates the highest level of health) - the Physical Component Score (PCS-12) and Mental Component Score (MCS-12). At times, the survey is also displayed via 8 domain scales that are also scored from 0 to 100 (where 100 indicates the highest level of health) as follows: Physical Function, Role Physical, Bodily Pain, General Health, Mental Health, Role Emotional, Social Function, and Vitality.
Patient derived outcome in terms of general quality of life, as determined by the SF-12 | 1 year post-operatively
  The 12-Item Short Form Health Survey (SF-12) is a patient reported outcome survey that evaluates functional health and well-being. The survey is converted into 2 summary measures that are scored from 0 to 100 (where 100 indicates the highest level of health) - the Physical Component Score (PCS-12) and Mental Component Score (MCS-12). At times, the survey is also displayed via 8 domain scales that are also scored from 0 to 100 (where 100 indicates the highest level of health) as follows: Physical Function, Role Physical, Bodily Pain, General Health, Mental Health, Role Emotional, Social Function, and Vitality.
Patient derived outcome in terms of general quality of life, as determined by the SF-12 | 3 years post-operatively
  The 12-Item Short Form Health Survey (SF-12) is a patient reported outcome survey that evaluates functional health and well-being. The survey is converted into 2 summary measures that are scored from 0 to 100 (where 100 indicates the highest level of health) - the Physical Component Score (PCS-12) and Mental Component Score (MCS-12). At times, the survey is also displayed via 8 domain scales that are also scored from 0 to 100 (where 100 indicates the highest level of health) as follows: Physical Function, Role Physical, Bodily Pain, General Health, Mental Health, Role Emotional, Social Function, and Vitality.
A survival analysis of the LCS Complete AP Glide knee prosthesis | 1 year post-operatively
  Kaplan Meier survivorship analysis estimates the proportion of a population that will survive past a certain time avoiding a certain event. In this study, the event is removal of any component for any reason, also known as revision for any reason. Survival estimates are provided when 40* devices are left still being followed.
A survival analysis of the LCS Complete AP Glide knee prosthesis | 3 years post-operatively
  Kaplan Meier survivorship analysis estimates the proportion of a population that will survive past a certain time avoiding a certain event. In this study, the event is removal of any component for any reason, also known as revision for any reason. Survival estimates are provided when 40* devices are left still being followed.
Assessment of component alignment and positioning | 3 months post-operatively
Assessment of component alignment and positioning | 1 year post-operatively
Assessment of component alignment and positioning | 3 years post-operatively
Assessment of radiolucencies | 3 months post-operatively
Assessment of radiolucencies | 1 year post-operatively
Assessment of radiolucencies | 3 years post-operatively
Assessment of Patella Tilt and patellofemoral alignment | 3 months, 1 yr, and 3 yrs

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Dong-A University medical centre, Pusan
  - Ewha Womans University Mokdong Hospital, Seoul
  - Severance Hospital, Yongsei University College of Medicine, Seoul